CLINICAL TRIAL: NCT00401778
Title: Trial of RAD001 in Patients With Operable Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Suresh S. Ramalingam, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024810
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2015-07-14 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-11

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): RAD001 5 mg/day for 21 days sequentially.
  Interventions: Drug: RAD001
- 3 (Active Comparator): RAD001 10 mg/day for 21 days sequentially.
  Interventions: Drug: RAD001
- Control (No Intervention): Patients who are eligible for the study but choose not to receive RAD001 treatment.

INTERVENTIONS:
Drug: RAD001 — Patients will be assigned to one of three treatment arms with RAD001 doses of 5, and 10 mg/day for 21-28 days sequentially taken orally in tablet form.
  Other Names: Everolimus
  Arms: 1; 3

SUMMARY:
This is a Phase 1b pre-operative lung cancer trial wherein patients with operable lung cancer will be treated with RAD001 to evaluate the target effects of this compounds on relevant molecular pathways and on the 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) uptake of the tumor by a positron emission tomography (PET) scan at baseline and immediately prior to surgery. The safety profile of RAD001 will also be evaluated.

DETAILED DESCRIPTION:
This is a Phase 1b pre-operative lung cancer trial wherein patients with operable lung cancer will be treated with RAD001 for 3-4 weeks to study the effects of the novel agent in relevant molecular pathways. The study will also assess the FDG uptake of the tumor at baseline and upon completion of therapy (before surgery) with a PET scan. The safety profile of RAD001 will also be evaluated.

New agents and regimens are urgently needed for lung cancer treatment. With the development of novel agents and small molecules designed to curtail the aggressive aspects of this disease, some progress has been realized. However, much more effort and insight will be required for further real gains to be made. We propose that studying the mammalian target of rapamycin (mTOR) axis, known to be abnormal in non-small cell lung cancer (NSCLC), and translating that knowledge into therapeutic adjustments can lead to meaningful advances in lung cancer treatment.

Approximately 35 patients will participate at Winship Cancer Institute of Emory University in Atlanta, Georgia.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed Stage I-IIIA non-small cell lung cancer (NSCLC) which is accessible to biopsy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Life-expectancy greater than 6 months.
* Adequate bone marrow, renal, hepatic, pulmonary and cardiac function as defined in the protocol.
* Patient must be at least 18 years of age.
* Must meet pre-entry requirements for timing of study parameters as specified in section 7.0.
* Female patients of child-bearing potential must have a negative serum pregnancy test within 48 hours of study initiation and be non-lactating.
* Patients of child-bearing potential must agree to use an effective form of contraception while on study and for 3 months following completion of study treatment.
* The use of granulocyte-colony stimulating factor (G-CSF) will be permitted in study participants.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Exclusion Criteria:

* Patient has received previous treatment for NSCLC.
* Known hypersensitivity to everolimus, sirolimus, or any of its excipients.
* Patient is pregnant or breast-feeding.
* Patient has incurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patient is unable to swallow RAD001 tablet.
* History of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of the malignancy being present within the past five years.
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80. Symptoms may include any reaction such as bronchospasm, generalized urticaria, systolic BP ≤ 80mm Hg, and angioedema.
* Final eligibility for a clinical trial is determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Ramalingam, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All enrolled patients were recruited through the multidisciplinary thoracic oncology clinics of Emory Clinic of Emory University.
Pre-assignment Details: Eligible patients were enrolled concurrently on the active and control arms. Patient preference for a specific arm was entertained until the control cohort was completely filled after which all patients were competitively enrolled on the active treatment arm of the study.
Groups:
- Control: No everolimus taken.
- Everolimus 5 mg: Everolimus dose of 5 mg/day for 21-28 days sequentially taken orally in tablet form.
- Everolimus 10 mg: Everolimus dose of 10 mg/day for 21-28 days sequentially taken orally in tablet form.
Period: Overall Study
Arm/Group | Control | Everolimus 5 mg | Everolimus 10 mg
Started | 10 | 12 | 11
Completed | 9 | 11 | 10
Not Completed | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Everolimus 5 mg | Everolimus 10 mg | Total
Number analyzed (Participants) | 10 | 12 | 11 | 33
Age, Continuous [Median (Full Range); unit: years] | 63 [54 to 77] | 58 [44 to 66] | 70 [35 to 75] | 64 [35 to 77]
Gender [Count of Participants; unit: Participants]
  Female | 6 | 6 | 7 | 19
  Male | 4 | 6 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 9
  White | 7 | 10 | 7 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response as Assessed Metabolically by Changes in Positron Emission Tomography (PET) Scan Between Baseline and Immediately Prior to Surgery.
Description: All patients had baseline imaging in a fasted state with 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18FDG)-PET scan and a repeat scan at 3 to 4 weeks later using routine clinical protocol for patient preparation, radiotracer administration and data acquisition. The repeat imaging occurred no longer than 24 hours before surgical resection.
Time Frame: Day 21
Measure: Number; unit: percentage of patients
Arm/Group | Control | Everolimus 5 mg | Everolimus 10 mg
Number analyzed (Participants) | 9 | 11 | 10
percentage of patients
  Stable metabolic disease (SMD) | 78 | 64 | 50
  Progressive metabolic disease (PM) | 22 | 36 | 50

2. Primary Outcome: Effects of RAD001 on the Regulation of Key Proteins Involved With the Mammalian Target of Rapamycin (mTOR) Axis in Tumor Specimens and Buccal Mucosa in Patients With Operable Non-small Cell Lung Cancer (NSCLC).
Description: Changes in the expression of key signaling proteins in the mTOR/phosphatidylinositol 3-kinase (PI3K) pathway were determined by immunohistochemistry using previously published protocols and manufacturers' recommendations for antigen retrieval and antibody dilution along with positive and negative controls. Two investigators assessed protein expression jointly by light microscopy. The degree of expression was assessed by intensity (0, 1+, 2+, 3+) and percentage of cell staining in line with published algorithm. A derivative score (immunoscore) ranging between 0 and 300 was calculated as the product of intensity and percent cell staining.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % change in immunoscore
Arm/Group | Control | Everolimus 5 mg | Everolimus 10 mg
Number analyzed (Participants) | 9 | 11 | 10
% change in immunoscore
  S6 | -36.06 (100.02) | -13.69 (144.05) | -77.03 (16.02)
  pS6 | -41.25 (65.62) | -61.57 (35.8) | -47.21 (44.96)
  pS6/S6 | -85.75 (20.15) | -100 (NA) — Insufficient tissue sample for testing | 128.57 (219.26)
  pMTOR | -6.58 (138.88) | 30 (153.95) | -63.82 (51.3)
  p4E-BP1 | -95.37 (4.24) | 150 (NA) — Insufficient tissue sample for testing | -78.75 (14.36)
  p70s6k | 25 (176.78) | 137.14 (442.07) | -78.62 (22.79)
  p70s6k Cytoplasmic | -19.17 (73.16) | 0.56 (14.93) | 305.37 (686.3)
  p70s6k Nuclear | -3.33 (100.17) | 135 (49.5) | 223.43 (437.7)
  pe1f4e | -50 (86.6) | 2.78 (5.56) | -27.13 (42.17)
  PAKT Nuclear | -33.33 (57.74) | NA (NA) — Insufficient tissue sample for testing | 0 (0)
  PAKT Cytoplasmic | 200 (469.04) | NA (NA) — Insufficient tissue sample for testing | -25 (50)
  Bim | -11.76 (NA) — Insufficient tissue sample for testing | NA (NA) — Insufficient tissue sample for testing | -21.76 (60.07)

3. Primary Outcome: Inhibition of Proliferation (Ki67) and Induction of Apoptosis (TUNEL Assay) in Tumor Specimens and Buccal Mucosa.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Safety and Tolerability of RAD001 as Pre-operative Therapy.
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Duration of Hospital Stay Following Surgery.
Time Frame: 6 months
Measure: Median (Full Range); unit: days
Groups:
- Everolimus 5 or 10 mg: Everolimus dose of 5 or 10 mg/day for 21-28 days sequentially taken orally in tablet form.
Arm/Group | Control | Everolimus 5 or 10 mg
Number analyzed (Participants) | 10 | 20
days | 5 [2 to 15] | 5 [3 to 43]

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- Everolimus 5 & 10 mg: Everolimus dose of 5 or 10 mg/day for 21-28 days sequentially taken orally in tablet form.
Arm/Group | Control | Everolimus 5 & 10 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/23
Other Adverse Events (participants affected / at risk) | 0/10 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=10) | Everolimus 5 & 10 mg (N=23)
Symptomatic Progression of Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 — One subject was enrolled to the study and was receiving RAD001 therapy. During week 2, she was hospitalized for symptomatic progression of her lung cancer.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=10) | Everolimus 5 & 10 mg (N=23)
Hyperglycemia (Blood and lymphatic system disorders) | 0 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Elevated Cholesterol (Vascular disorders) | 0 | 13
Fatigue (General disorders) | 0 | 14
Diarrhea (Gastrointestinal disorders) | 0 | 3
Night Sweats (General disorders) | 0 | 3
Fever (General disorders) | 0 | 3
Elevated Creatinine (Renal and urinary disorders) | 0 | 8
Insomnia (General disorders) | 0 | 5
Hoarseness (General disorders) | 0 | 2
Heartburn (Gastrointestinal disorders) | 0 | 2
Weight-loss (Metabolism and nutrition disorders) | 0 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Nausea (General disorders) | 0 | 8
Elevated ALT (Blood and lymphatic system disorders) | 0 | 9
Elevated AST (Blood and lymphatic system disorders) | 0 | 10
Elevated Alkaline Phosphatase (Blood and lymphatic system disorders) | 0 | 9
Hypocalcemia (Blood and lymphatic system disorders) | 0 | 12
Hyponatremia (Blood and lymphatic system disorders) | 0 | 10
Hypokalemia (Blood and lymphatic system disorders) | 0 | 10
Anemia (Blood and lymphatic system disorders) | 0 | 12
Hypophosphatemia (Blood and lymphatic system disorders) | 0 | 4
Hypoalbuminemia (Blood and lymphatic system disorders) | 0 | 12
Vertigo (Ear and labyrinth disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Difficulty in Breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertriglyceridemia (Blood and lymphatic system disorders) | 0 | 15
Headache (Nervous system disorders) | 0 | 3
Low Leukocytes (Immune system disorders) | 0 | 3
Mouth Sores (Skin and subcutaneous tissue disorders) | 0 | 5
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Bronchitis (Infections and infestations) | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Reflux (Gastrointestinal disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Burning with Urination (Renal and urinary disorders) | 0 | 1
Pain in Lower Flank (General disorders) | 0 | 1
Intermittent Discomfort in Left Leg (General disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Low Platelets (Blood and lymphatic system disorders) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
MRSA Bacteremia (Infections and infestations) | 0 | 1
Acute Renal Failure (Renal and urinary disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 7
Upper Respiratory Infection (Infections and infestations) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Edema (Blood and lymphatic system disorders) | 0 | 5
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Sinusitis (Musculoskeletal and connective tissue disorders) | 0 | 5
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain (Nervous system disorders) | 0 | 6
Neuropathy (Nervous system disorders) | 0 | 2
Dizziness (General disorders) | 0 | 2
Restlessness (General disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Confusion (General disorders) | 0 | 1
Loss of Energy (General disorders) | 0 | 1
Difficulty in Walking (General disorders) | 0 | 1
Loss of Balance (General disorders) | 0 | 1
Hot Flashes (Endocrine disorders) | 0 | 1
Hypercalcemia (Blood and lymphatic system disorders) | 0 | 1
Conjuctivitis (Eye disorders) | 0 | 1
Photosensitivity (General disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Ear Ache (Ear and labyrinth disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 0 | 1
Cramping Feet (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes